CLINICAL TRIAL: NCT05286099
Title: The Surveillance of Development and Progression of Hepatocellular Carcinoma
Brief Title: The Surveillance of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chinese PLA General Hospital, Chinese PLA General Hospital
Other Study IDs: S2022-001
Record Dates: First submitted 2022-02-22; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Imaging examination and/or blood test — Imaging examination and/or blood test will be performed at a certain time

SUMMARY:
Early detection of hepatocellular carcinoma is vita to the prognosis of patient. In this study, the occurrence and development of liver cancer were supervised by imaging examination, and the dysplastic nodules will be distinguished from early hepatocellular carcinoma through macro-imaging and micro-pathological features.

ELIGIBILITY:
Inclusion Criteria:

- Patients with Hepatitis B and cirrhosis Accept regular imaging examination. Pathological diagnosis of liver cancer.

Exclusion Criteria:

- Can't tolerate the enhanced imaging examination Poor medical compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatitis B, liver cirrhosis, or atypical hyperplasia nodules confirmed or suspected by enhanced imaging examination will be enrolled, the contrast-enhanced ultrasound and/or enhanced magnetic resonance imaging will be performed every three months or half a year to observe the size and contrast-enhanced features of the nodules. If the size or enhancement features change, there will a puncture biopsy under the guidance of ultrasound, and if malignant tumor cells are found, the follow-up will be terminated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Effective detection of early hepatocellular carcinoma | 2 years
  The occurrence of early hepatocellular carcinoma

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chinese PLA general hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided